CLINICAL TRIAL: NCT03986541
Title: Association Between Tumour Amphiregulin, Epiregulin and Epidermal Growth Factor Receptor (EGFR) Expression and Response to Anti-EGFR Agents in Colorectal Cancer
Brief Title: AREG, EREG and EGFR: Response to Anti-EGFR Agents in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: University of Liverpool (Other); University of Manchester (Other); Newcastle University (Other); University of Nottingham (Other); University of Sheffield (Other)
Responsible Party: Principal Investigator, Philip Quirke, Professor Philip Quirke, University of Leeds
Other Study IDs: N6AREG/EREG
Record Dates: First submitted 2019-06-13; First posted 2019-06-14 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer Stage IV
Keywords: colorectal cancer; anti-EGFR agents; cetuximab; panitumumab; amphiregulin; epiregulin; EGFR
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Consent sought for retention of pathological specimens of colorectal cancer for future Research Ethics Committee approved bowel cancer research (not a prerequisite to study participation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: Patients with advanced colorectal cancer previously treated with an anti-EGFR agent (panitumumab or cetuximab).
  Interventions: Diagnostic Test: Immunohistochemistry
- Prospective cohort: Patients with advanced colorectal cancer newly starting treatment with an anti-EGFR agent (panitumumab or cetuximab).
  Interventions: Diagnostic Test: Immunohistochemistry

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry — Assessment of tumour amphiregulin, epiregulin and EGFR expression by immunohistochemistry.

SUMMARY:
Observational study investigating the relationship between tumour amphiregulin, epiregulin and epithelial growth factor receptor expression and response to anti-EGFR agents in advanced colorectal cancer.

DETAILED DESCRIPTION:
Background:

The anti-EGFR agents, cetuximab and panitumumab are approved by NICE for the first-line treatment of patients with RAS wild-type (RAS-wt) advanced colorectal cancer (aCRC). However RAS-wt status is not sufficient to guarantee anti-EGFR benefit. Differential tumour expression of the EGFR ligands, amphiregulin (AREG) and epiregulin (EREG), as well as the EGFR receptor itself, are putative predictive biomarkers for response to anti-EGFR agents and may therefore help better identify patients who will benefit from treatment.

Objectives:

This study aims to assess the utility of tumour AREG, EREG and/or EGFR expression, alone or in combination, as predictive biomarkers for response to anti-EGFR agents in aCRC. The investigators will develop a scoring system and categorical cut off points to differentiate AREG/EREG/EGFR positive and negative cases and correlate these with response to therapy as assessed by:

Primary endpoint: Progression Free Survival (PFS) Secondary endpoints: Overall Survival (OS), Objective Response Rate (ORR), Disease Control Rate (DCR) Finally, the investigators will utilise digital pathology and artificial intelligence (AI) technologies to automate as far as possible the process of evaluating AREG/EREG/EGFR status.

During the study, the investigators will monitor the costs of implementing the test and time taken to derive test results in order to facilitate cost-effectiveness calculations and assess the feasibility of delivering the test in future routine clinical practice.

Study Design:

A multicentre UK observational cohort study (retrospective and prospectively recruited cohorts).

Study population:

Patients with RAS-wt aCRC who received or are receiving standard care palliative treatment with an anti-EGFR agent and chemotherapy of physician's choice. Within the retrospective cohort, patients who received single agent anti-EGFR therapy under previous Cancer Drugs Fund criteria will be accepted.

Key Inclusion Criteria:

* Biopsy proven advanced colorectal adenocarcinoma at time treatment commenced (either inoperable metastatic disease at diagnosis or inoperable recurrent disease)
* Aged 18 or over at time treatment commenced
* The patient has received or has consented to receive treatment with cetuximab or panitumumab

Key Exclusion Criteria:

* Stage I, II or III colorectal adenocarcinoma
* RAS mutant disease
* Eligible for potentially curative surgery (prospective cohort)
* Underwent cancer surgery subsequent to anti-EGFR therapy (retrospective cohort)
* Unable to provide informed consent (with the exception of patients in the retrospective cohort who have passed away)

Procedures:

The study is observational and does not involve participants undergoing any study-specific investigations or treatments. Results of routine investigations and outcomes from standard care with an anti-EGFR agent will be collected from medical notes and, for the prospective cohort, during routine clinic appointments. Date of death will also be recorded. Initial and follow-up radiological and clinical assessments will occur as per local standard practice. Previously obtained pathological specimens will be retrieved for immunohistochemical analysis of tumour AREG, EREG and EGFR expression.

Treatment During Study:

This study will observe outcomes from standard first line palliative treatment of RAS-wt aCRC. In line with current NICE guidelines, such treatment will involve physician's choice of panitumumab or cetuximab in combination with:

* 5-fluorouracil, folinic acid and oxaliplatin (FOLFOX) or
* 5-fluorouracil, folinic acid and irinotecan (FOLFIRI) Where RAS mutation status is only available after commencement of treatment and the anti-EGFR agent is therefore commenced in cycle two, patients may still be recruited to the study.

It is anticipated that most patients in the retrospective cohort will have received current standard first line palliative treatment of RAS-wt aCRC as above. However, patients who were treated with single agent anti-EGFR therapy under previous Cancer Drugs Fund criteria may still be recruited.

Statistical Methods:

Sample size:

Data from 480 patients will be collected for the retrospective cohort and 480 patients will be recruited to the prospective cohort.

Primary endpoint analysis:

PFS will be calculated from date of commencing treatment to date of progression or death from any cause (whichever is sooner). Time of progression will be determined clinically or radiologically by the participant's treating oncologist. Where the anti-EGFR agent was commenced in cycle 2, the definition of the start of treatment will remain cycle 1 day 1 of palliative chemotherapy.

Key secondary endpoint analyses:

OS will be determined from date of commencing treatment to death. ORR is the proportion of patients with documented radiological complete or partial response on first follow-up imaging whereas DCR is the proportion of patients with either radiologically stable disease or a response. For the purpose of these analyses, those without follow-up imaging will be assumed to have progressed.

AREG/EREG/EGFR expression will be assessed as a continuous variable and using dichotomous classifiers ('high' and 'low') for each marker individually and in combination. Subgroup analyses will be performed for BRAF mutation positive tumours, primary tumour location (right versus left colon, and rectum) and previous surgery (primary excised versus in situ). Within the retrospective cohort, those who received single agent anti-EGFR therapy under previous Cancer Drugs Fund criteria will be analysed separately.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven advanced colorectal adenocarcinoma at time treatment commenced (either inoperable metastatic disease at diagnosis or inoperable recurrent disease)
* Aged 18 or over at time treatment commenced
* The patient has received or has consented to receive treatment with cetuximab or panitumumab

Exclusion Criteria:

* Stage I, II or III colorectal adenocarcinoma
* RAS mutant disease
* Eligible for potentially curative surgery (prospective cohort)
* Underwent cancer surgery subsequent to anti-EGFR therapy (retrospective cohort)
* Unable to provide informed consent (with the exception of patients in the retrospective cohort who have passed away)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RAS-wt aCRC who received or are receiving standard care palliative treatment with an anti-EGFR agent and chemotherapy of physician's choice. Within the retrospective cohort, patients who received single agent anti-EGFR therapy under previous Cancer Drugs Fund criteria will be accepted.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Progression free survival | March 2023
  PFS will be calculated from date of commencing treatment to date of progression or death from any cause (whichever is sooner). Time of progression will be determined clinically or radiologically by the participant's treating oncologist.

SECONDARY OUTCOMES:
Overall survival | March 2023
  OS will be determined from date of commencing treatment to death.
Objective response rate | 8-12 weeks post commencement of treatment
  ORR is the proportion of patients with documented radiological complete or partial response on first follow-up imaging.
Disease control rate | 8-12 weeks post commencement of treatment
  DCR is the proportion of patients with either radiologically stable disease or a response on first follow-up imaging

CONTACTS AND LOCATIONS:
Overall Officials: Philip Quirke, PhD FRCPath, Principal Investigator — University of Leeds - Institute of Medical Research at St James's
Locations (7):
- United Kingdom (7):
  - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield, West Yorkshire
  - St James's University Hospital, Leeds
  - The Christie NHS Foundation Trust, Manchester
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No